CLINICAL TRIAL: NCT03587766
Title: Phase 2 Randomized, Multicenter, Double-blinded Safety and Efficacy Study to Evaluate Oral Fexinidazole Dosing Regimens for the Treatment of Adult Patients With Chronic Indeterminate Chagas Disease
Brief Title: Oral Fexinidazole Dosing Regimens for the Treatment of Adults With Chronic Indeterminate Chagas Disease
Acronym: FEXI12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNDi-FEX-12-CH; 2016-004905-15 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-07-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Chagas' Disease (Chronic) Nos
Keywords: Trypanosoma cruzi Infection; Chagas' Disease; Trypanosomiasis, South American; American Trypanosomiasis; Kissing bug
MeSH Terms: conditions — Chagas Disease; Bronchiolitis Obliterans Syndrome; Pyloric Stenosis, Hypertrophic | interventions — fexinidazole

STUDY DESIGN:
Intervention Model Description: This study is designed as a double-blind, randomized, prospective, comparative, pharmacokinetic-pharmacodynamic, and proof-of-concept trial design, with three-parallel groups and historical placebo control in patients with chronic indeterminate Chagas Disease.
Who Masked: Participant, Investigator
Masking Description: As the study is double-blinded, the patient, investigators, pharmacist(s) and DNDi study team members involved with the clinical trial implementation will remain blinded to treatment allocation for the duration of the clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Fexinidazole (FEXI) 600 mg x 10 days in a single daily dose orally (1 fexinidazole 600 mg tablet and 1 fexinidazole matching placebo oral tablet administered in a single daily dose) (total dose: 6.0 g).
  Interventions: Drug: Fexinidazole; Drug: Placebo Oral Tablet
- Group B (Experimental): Fexinidazole (FEXI) 1200 mg x 3 days orally (2 fexinidazole 600 mg tablets administered in a single daily dose for 3 days), to be followed by matching placebo oral tablet for 7 days (2 fexinidazole matching placebo oral tablets administered once daily for 7 days) (total dose: 3.6 g).
  Interventions: Drug: Fexinidazole; Drug: Placebo Oral Tablet
- Group C (Experimental): Fexinidazole (FEXI) 600 mg for 3 days, followed by 1200 mg in a single daily dose orally for 4 days (1 fexinidazole 600 mg tablet AND 1 fexinidazole matching placebo oral tablet administered in a single daily dose for 3 days, to be followed by 2 fexinidazole 600 mg tablets for 4 days), then followed by matching placebo oral tablet for 3 days (2 fexinidazole matching placebo tablets administered once daily for 3 days) (total dose: 6.6 g).
  Interventions: Drug: Fexinidazole; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Fexinidazole — Drug: fexinidazole (FEXI)
  Other Names: FEXI
Drug: Placebo Oral Tablet — Drug: fexinidazole
  Other Names: Placebo

SUMMARY:
This study focuses on the evaluation of low doses (600 and 1200 mg) and short treatment duration (at 3, 7 and 10 days) of fexinidazole (Fexi) to determine the minimal efficacious and safe dose for the treatment of adult patients with chronic indeterminate Chagas Disease (CD).

DETAILED DESCRIPTION:
Fexi anti-protozoal activity against T. cruzi has been demonstrated by various in vitro and in vivo studies.

Patients will be randomly assigned to receive one of three different treatment regimen arms containing either the active drug or matching placebo tablet

Following conclusion of 12 months of follow-up of DNDi-CH-FEXI-001 clinical trial, unblinded data review showed high sustained parasite clearance rates of FEXI even at the lowest dose tested (1200 mg 2 weeks), including in patients that received < 3days treatment.

ELIGIBILITY:
Screening Criteria:

* Signed, written informed consent form
* Age >18 to < 60 years
* Weight > 50 kg to < 90 kg
* Diagnosis of T. cruzi infection by:
* Conventional serology (a minimum of two positive tests [Conventional ELISA, Recombinant Elisa, Chemiluminescence Immunoassays and/or Indirect Immunofluorescence (IIF)]
* Ability to comply with all protocol specified tests and visits and have a permanent address
* No signs and/or symptoms of the chronic cardiac and/or digestive form of Chagas Disease (CD) (as per study operating procedures)
* No personal history of mental disability or suicidal tendencies
* No acute or chronic health conditions, that in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the trial drug (such as acute infections, history of HIV infection, liver, and renal disease requiring treatment)
* No formal contraindication to FEXI (according to the latest available Investigator's Brochure)
* No history of hypersensitivity, allergic, or serious adverse reactions to any of the "nitro-imidazoles" compound, and/or its components
* No history of CD treatment with BZN, FEXI or Nifurtimox (NFX) at any time in the past
* No history of alcohol abuse or any other drug addiction (as per Study Manual of Operations)
* No condition that prevents patient from taking oral medication
* No concomitant medication with drug known risk of Torsade de Pointe, according AZCERT Scientific Publications and Sudden Arrhythmia Death Syndromes Foundation (SADS Foundation) (https://www.crediblemeds.org/index.php/new-drug-list)
* No family history of sudden death
* No family history of sudden infant death syndrome

Inclusion Criteria:

Following the screening period, patients must also meet all of the following inclusion criteria to be eligible for randomization:

* Confirmed diagnosis of T. cruzi infection by:
* Serial qualitative PCR (three samples collected over a single day, at least one of which must be positive),

and

* Conventional serology (a minimum of two positive tests must be positive, Conventional ELISA, Recombinant Elisa, Chemiluminescence immunoassays and/or IIF)
* Women in reproductive age must have a negative serum pregnancy test at screening, must not be breastfeeding, must consistently use a highly effective contraceptive method until end of treatment and estimated FEXI, M1 and M2 clearance (total of 21 days). After this, contraception is no longer required.
* Normal ECG (Heart rate: 50-100bpm; PR interval ≤200 msec, QRS complex ≤120 msec, and QT interval corrected for heart rate (QTc) ≥350msec and ≤450 msec interval durations) at screening
* 24 hour Holter-monitoring with no clinically relevant arrythmias (defined as Ventricular Tachycardia (defined as >3 ventricular beats with >100bpm); Sustained Accelerated Idio-Ventricular rhythm (defined as >30 seconds duration and Heart Rate (HR): 50bpm<HR<100bpm); frequent Ventricular Premature Beats (10/hour); Atrial Fibrillation/flutter; Mobitz type 2 second degree AV block; High degree and complete AV block; Bradycardia episodes <40bpm)

Exclusion Criteria:

* Signs and/or symptoms of chronic cardiac and/or digestive form of CD (as per Study Manual of Operations).
* History of cardiomyopathy, heart failure, or ventricular arrhythmia.
* History of digestive surgery or mega syndromes.
* Personal history of mental disability or suicidal tendencies
* Hospital Anxiety and Depression Scale (HADS - Appendix 1) self-assessment score >11 in each of the sub-scales. (Note: If HADS score >11, retesting would be allowed before after a minimum period of 15 days and referral to counseling/evaluation.)
* Any other acute or chronic health conditions that, in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the trial drug (such as acute infections, history of HIV infection, diabetes, uncontrolled systolic/diastolic blood pressure, liver, and renal diseases requiring medical treatment).
* Laboratory test values considered clinically significant or out of the allowable range at selection period as follows:

  * Total White Blood Count (WBC) must be within the normal range, with an acceptable margin of +/- 5% (3,800 - 10,500 / mm3).
  * Platelets must be within the normal range up to 550,000/mm3
  * Total bilirubin must be within the normal range
  * Transaminases (ALT and AST) must be within the normal range, with an acceptable margin of 25% above the upper limit of normality (ULN), < 1.25 x ULN.
  * Creatinine must be within an acceptable margin of 10% above the ULN, <1.10 x ULN.
  * Alkaline phosphatase must be within the normal range up to Grade 1 CTCAE (<,2.5 x ULN)
  * Gamma-glutamyl Transpeptidase (GGT) must be within the normal range up to 2x ULN.
  * Fasting glucose (minimum of 8 hours from latest meal) must be within the normal range
  * Electrolytes (Ca, Mg, K) must be within the normal range
  * Hepatitis screen must be negative for acute and/or chronic infection (Hepatitis A antibody, Imunoglobulina M (IgM); Hepatitis B surface Ag, Hepatitis B

If the results of the blood tests (hematology and biochemistry) are out of the ranges defined above, but within the limits of CTCAE (version 4.03) Grade 1, and this laboratory finding is considered as non-clinically significant, a new sample can be collected for a retest. Only one retest will be allowed within the screening period.

If the result of the retest is within the margins defined above, the Investigator will review the parameter(s) together with all other medical information available (medical history, clinical examinations, vital signs, etc.) and upon his/her medical judgement will decide if the patient is eligible or not for trial randomization.

Any condition that prevents the patient from taking oral medication.

* Patients with any contra-indication (known hypersensitivity) to any nitroimidazoles, e.g. metronidazole
* Patients with history of allergy (serious or not), allergic skin rash, asthma, intolerance, sensitivity or photosensitivity to any drug
* Any concomitant use of allopurinol, antimicrobial, anti-parasitic agents, and/or of herbal medicines, food supplements and energetic drinks
* Any concomitant medication with drug known risk of Torsade de Pointe, according AZCERT Scientific Publications and SADS Foundation (www.crediblemeds.org/index.php/new-drug-list)
* Any planned surgery likely to interfere with the trial conduction and/or treatment evaluation
* Unlikely to return for study visits, comply with study treatment and co-operate with the trial-related procedures.
* Any previous participation in any clinical trial for Chagas Disease treatment evaluation
* Participation in another trial at the same time or within 3 months prior to selection (according to local regulations).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | 12 months

SECONDARY OUTCOMES:
Pharmacokinetic : measure of blood concentration of fexinidazole, fexinidazole sulfoxide and fexinidazole sulfone in order to determine AUC0-t values, for all dose levels. | D0 (pre-dose), Day 1, Day 2, Day 3, and at steady-state phase (week 2-10).
Pharmacokinetic : measure of blood concentration of fexinidazole, fexinidazole sulfoxide and fexinidazole sulfone in order to determine Cmax values, for all dose levels. | D0 (pre-dose), Day 1, Day 2, Day 3, and at steady-state phase (week 2-10).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Gascón, MD, Principal Investigator — Centro de Salud Internacional, Hospital Clínico de Barcelona ISGlobal - Barcelona Institute for Global Health
Locations (1):
- Hospital Clinic, Barcelona, Catalunia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Not yet decided how Individual Participant Data (IPD) will be shared, This action is under internal review within DNDi.

REFERENCES:
- [Background] WHO | Chagas disease (American trypanosomiasis) [Internet]. WHO. [cited 2013 Aug 22]. Available from: http://www.who.int/mediacentre/factsheets/fs340/en/index.html
- [Background] Bern C, Montgomery SP. An estimate of the burden of Chagas disease in the United States. Clin Infect Dis. 2009 Sep 1;49(5):e52-4. doi: 10.1086/605091. PMID 19640226
- [Background] Torreele E, Bourdin Trunz B, Tweats D, Kaiser M, Brun R, Mazue G, Bray MA, Pecoul B. Fexinidazole--a new oral nitroimidazole drug candidate entering clinical development for the treatment of sleeping sickness. PLoS Negl Trop Dis. 2010 Dec 21;4(12):e923. doi: 10.1371/journal.pntd.0000923. PMID 21200426
- [Background] Raether W, Seidenath H. The activity of fexinidazole (HOE 239) against experimental infections with Trypanosoma cruzi, trichomonads and Entamoeba histolytica. Ann Trop Med Parasitol. 1983 Feb;77(1):13-26. doi: 10.1080/00034983.1983.11811668. PMID 6411009
- [Background] Moraes CB, Giardini MA, Kim H, Franco CH, Araujo-Junior AM, Schenkman S, Chatelain E, Freitas-Junior LH. Nitroheterocyclic compounds are more efficacious than CYP51 inhibitors against Trypanosoma cruzi: implications for Chagas disease drug discovery and development. Sci Rep. 2014 Apr 16;4:4703. doi: 10.1038/srep04703. PMID 24736467
- [Background] Bahia MT, de Andrade IM, Martins TA, do Nascimento AF, Diniz Lde F, Caldas IS, Talvani A, Trunz BB, Torreele E, Ribeiro I. Fexinidazole: a potential new drug candidate for Chagas disease. PLoS Negl Trop Dis. 2012;6(11):e1870. doi: 10.1371/journal.pntd.0001870. Epub 2012 Nov 1. PMID 23133682
- [Background] Caldas S, Caldas IS, Cecilio AB, Diniz LF, Talvani A, Ribeiro I, Bahia MT. Therapeutic responses to different anti-Trypanosoma cruzi drugs in experimental infection by benznidazole-resistant parasite stock. Parasitology. 2014 Oct;141(12):1628-1637. doi: 10.1017/S0031182014000882. PMID 25045804
- [Background] Munoz J, Gomez i Prat J, Gallego M, Gimeno F, Trevino B, Lopez-Chejade P, Ribera O, Molina L, Sanz S, Pinazo MJ, Riera C, Posada EJ, Sanz G, Portus M, Gascon J. Clinical profile of Trypanosoma cruzi infection in a non-endemic setting: immigration and Chagas disease in Barcelona (Spain). Acta Trop. 2009 Jul;111(1):51-5. doi: 10.1016/j.actatropica.2009.02.005. Epub 2009 Mar 5. PMID 19426663
- [Background] Rodriques Coura J, de Castro SL. A critical review on Chagas disease chemotherapy. Mem Inst Oswaldo Cruz. 2002 Jan;97(1):3-24. doi: 10.1590/s0074-02762002000100001. PMID 11992141
- [Background] Rassi A Jr, Rassi A, Marin-Neto JA. Chagas disease. Lancet. 2010 Apr 17;375(9723):1388-402. doi: 10.1016/S0140-6736(10)60061-X. PMID 20399979
- [Background] Pinto Dias JC. The treatment of Chagas disease (South American trypanosomiasis). Ann Intern Med. 2006 May 16;144(10):772-4. doi: 10.7326/0003-4819-144-10-200605160-00012. No abstract available. PMID 16702594
- [Background] Castro AM, Luquetti AO, Rassi A, Rassi GG, Chiari E, Galvao LM. Blood culture and polymerase chain reaction for the diagnosis of the chronic phase of human infection with Trypanosoma cruzi. Parasitol Res. 2002 Oct;88(10):894-900. doi: 10.1007/s00436-002-0679-3. Epub 2002 Jun 15. PMID 12209329
- [Background] de Castro AM, Luquetti AO, Rassi A, Chiari E, Galvao LM. Detection of parasitemia profiles by blood culture after treatment of human chronic Trypanosoma cruzi infection. Parasitol Res. 2006 Sep;99(4):379-83. doi: 10.1007/s00436-006-0172-5. Epub 2006 Mar 29. PMID 16570199
- [Background] Britto C, Cardoso MA, Vanni CM, Hasslocher-Moreno A, Xavier SS, Oelemann W, Santoro A, Pirmez C, Morel CM, Wincker P. Polymerase chain reaction detection of Trypanosoma cruzi in human blood samples as a tool for diagnosis and treatment evaluation. Parasitology. 1995 Apr;110 ( Pt 3):241-7. doi: 10.1017/s0031182000080823. PMID 7724232
- [Background] Solari A, Ortiz S, Soto A, Arancibia C, Campillay R, Contreras M, Salinas P, Rojas A, Schenone H. Treatment of Trypanosoma cruzi-infected children with nifurtimox: a 3 year follow-up by PCR. J Antimicrob Chemother. 2001 Oct;48(4):515-9. doi: 10.1093/jac/48.4.515. PMID 11581230
- [Background] Galvao LM, Chiari E, Macedo AM, Luquetti AO, Silva SA, Andrade AL. PCR assay for monitoring Trypanosoma cruzi parasitemia in childhood after specific chemotherapy. J Clin Microbiol. 2003 Nov;41(11):5066-70. doi: 10.1128/JCM.41.11.5066-5070.2003. PMID 14605140
- [Background] Schijman AG, Altcheh J, Burgos JM, Biancardi M, Bisio M, Levin MJ, Freilij H. Aetiological treatment of congenital Chagas' disease diagnosed and monitored by the polymerase chain reaction. J Antimicrob Chemother. 2003 Sep;52(3):441-9. doi: 10.1093/jac/dkg338. Epub 2003 Aug 13. PMID 12917253
- [Background] Flores-Chavez M, Bosseno MF, Bastrenta B, Dalenz JL, Hontebeyrie M, Revollo S, Breniere SF. Polymerase chain reaction detection and serologic follow-up after treatment with benznidazole in Bolivian children infected with a natural mixture of Trypanosoma cruzi I and II. Am J Trop Med Hyg. 2006 Sep;75(3):497-501. PMID 16968928
- [Background] Duffy T, Bisio M, Altcheh J, Burgos JM, Diez M, Levin MJ, Favaloro RR, Freilij H, Schijman AG. Accurate real-time PCR strategy for monitoring bloodstream parasitic loads in chagas disease patients. PLoS Negl Trop Dis. 2009;3(4):e419. doi: 10.1371/journal.pntd.0000419. Epub 2009 Apr 21. PMID 19381287
- [Background] Ramirez JD, Guhl F, Umezawa ES, Morillo CA, Rosas F, Marin-Neto JA, Restrepo S. Evaluation of adult chronic Chagas' heart disease diagnosis by molecular and serological methods. J Clin Microbiol. 2009 Dec;47(12):3945-51. doi: 10.1128/JCM.01601-09. Epub 2009 Oct 21. PMID 19846646
- [Background] Diez M, Favaloro L, Bertolotti A, Burgos JM, Vigliano C, Lastra MP, Levin MJ, Arnedo A, Nagel C, Schijman AG, Favaloro RR. Usefulness of PCR strategies for early diagnosis of Chagas' disease reactivation and treatment follow-up in heart transplantation. Am J Transplant. 2007 Jun;7(6):1633-40. doi: 10.1111/j.1600-6143.2007.01820.x. PMID 17511688
- [Derived] Pinazo MJ, Forsyth C, Losada I, Esteban ET, Garcia-Rodriguez M, Villegas ML, Molina I, Crespillo-Andujar C, Gallego M, Ballart C, Ramirez JC, Aden T, Hoerauf A, Pfarr K, Vaillant M, Marques T, Fernandes J, Blum B, Ribeiro I, Sosa-Estani S, Barreira F, Gascon J; FEXI-12 Study Team. Efficacy and safety of fexinidazole for treatment of chronic indeterminate Chagas disease (FEXI-12): a multicentre, randomised, double-blind, phase 2 trial. Lancet Infect Dis. 2024 Apr;24(4):395-403. doi: 10.1016/S1473-3099(23)00651-5. Epub 2024 Jan 11. PMID 38218194